CLINICAL TRIAL: NCT05335343
Title: Evaluation of the Relationship Between Healthy Eating and Intrinsic Capacity in Elderly Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: HEICITY
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Healthy Eating Index; Muscle Strain; Frailty
Keywords: healthy eating; intrinsic capacity; elderly
MeSH Terms: conditions — Sprains and Strains; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The aim of this study is to evaluate the relationship between intrinsic capacity and healthy eating in elderly individuals.

DETAILED DESCRIPTION:
The relationship between the healthy eating index and intrinsic capacity in elderly individuals is unknown.

The aim of this study is to evaluate the relationship between intrinsic capacity and healthy eating in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Those who agreed to participate in the study
* Orally fed

Exclusion Criteria:

* Not voluntarily participating in the research
* Having a serious life-threatening condition (critical illness, hospitalization in the intensive care unit, acute complication)
* Those who do not have a mental disability that cannot answer the questions (Mental retardation, Alzheimer's, etc.)
* Major psychiatric illness
* congenital or acquired muscle disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals over the age of 65
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between intrinsic capacity and healthy eating | 2 week
  Relationship between intrinsic capacity and healthy eating

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Abdülhamid Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided